CLINICAL TRIAL: NCT05875779
Title: Developing Vaccine Educators Within Practices of Community Healthcare Providers: a Pragmatic, Randomized Controlled Trial of Peer Education to Promote Vaccine Acceptance
Brief Title: Peer Education as a Strategy to Promote Vaccine Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-01526
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Vaccine Acceptance
Keywords: Vaccine confidence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-led vaccine education intervention (Experimental): Parents randomized to peer-led vaccine education intervention.
  Interventions: Behavioral: Peer-led vaccine education intervention
- Usual Care (No Intervention): Parents randomized to usual care.

INTERVENTIONS:
Behavioral: Peer-led vaccine education intervention — The intervention will be delivered face-to-face by a trained peer-educator and will consist of one session of 10-20 minutes.
  Peer vaccine educators will receive written vaccine materials for distribution. These materials will present content that accurately represents the risks and benefits of vaccination.
  Responsibilities of the vaccine educators will be to: provide motivational interviewing with patients, provide vaccine counseling, address questions and concerns regarding available vaccines, brief clinical provider on hesitant patients and areas of their vaccine-related concerns, and provide follow-up with participants at day 30, day 60 and day 90 for additional engagement.
  Arms: Peer-led vaccine education intervention

SUMMARY:
Effective interventions to improve uptake of vaccines among hesitant groups are urgently needed. Peer education is an effective intervention in modifying health behaviors in other conditions and may be effective in promoting vaccine confidence but has not been studied. To fill this knowledge gap, we will enroll approximately 152 parents of children age 0-18 months who are eligible for pneumococcal conjugate (PCV-13) vaccine and randomize them 1:1 to a peer-led vaccine education intervention or usual care.

ELIGIBILITY:
Inclusion Criteria:

1. A parent of a child aged 0 to 18 months born at ≥35 weeks' gestation who is eligible for a dose of PCV-13. Eligibility by age defined as follows:

   1. Age 0-6 months: never received first dose or is >8 weeks from last dose (3 doses scheduled in this age group at 2, 4, and 6 months)
   2. Age 7-11 months: never received first dose or is > 8 weeks from last dose (2 doses scheduled in this age group if started at 7 months)
   3. 12-18 months: never received first dose, is >8 weeks from last dose (2 doses scheduled in this age group if started at 12 months) or is due for booster at 12-18 months having received primary series between age 2-11 months.
2. Self-identifies as Orthodox Jewish.
3. Is able to provide informed consent.

Exclusion Criteria:

1. Unable to communicate verbally in English or Yiddish
2. Unwilling or unable to utilize a Yiddish in-person or telephone interpreter
3. Has already participated in this study as an eligible adult or parent. A parent will only be able to participate in this study once (i.e. for only one child in the family that is eligible)
4. Has an appointment at clinic that day to specifically receive vaccines.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Ages 0 Months to 18 Months at Enrollment who Receive at least One Dose of PCV-13 Vaccine by 3 Months Post-Enrollment | Month 3 Post-Enrollment
  Outcome will be determined via review of patient medical chart.

SECONDARY OUTCOMES:
Number of Participants Ages 1 Month to 18 Months at Enrollment who Receive at least One Dose of PCV-13 Vaccine by 1 Month Post-Enrollment | Month 1 Post-Enrollment
  Outcome will be determined via review of patient medical chart.
Percentage of Days Under-immunized at 3 Months among Participants Ages 0 Months to 18 Months at Enrollment | Month 1 Post-Enrollment
  To obtain the percentage of days underimmunized, investigators will sum the days late across all 4 doses of PCV-13 doses and will divide this by the maximum cumulative number of days a child could be late if they had received no vaccine doses by their age one month post study enrollment. If a dose was never received, the maximum number of days late a child could be for dose will be: age at enrollment in days+31 days minus the latest age in days in which that dose should have been received.

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Carmody, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Grossman School of Medicine, Division of Infectious Diseases, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Ellie Carmody, MD, ellie.carmody@nyulangone.org.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to ellie.carmody@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hoffman E, Kahan T, Auerbach E, Brody H, Abramson NN, Haiken S, Shields D, Elyasi A, Ifrah S, Frenkel-Schick A, Zyskind I, Knoll M, Carmody E. Peer education as a strategy to promote vaccine acceptance: A randomized controlled trial within New York community healthcare practices. Vaccine. 2024 Nov 14;42 Suppl 5:126028. doi: 10.1016/j.vaccine.2024.05.076. Epub 2024 Jun 10. PMID 38862308